CLINICAL TRIAL: NCT04743505
Title: Phase I/II Study Exploring the Safety and Efficacy of Combining APL-101 With Frontline Osimertinib in Patients With EGFR-mutated Metastatic Non-small Cell Lung Cancer (NSCLC)
Brief Title: Safety and Efficacy of Combining APL-101 With Frontline Osimertinib in Patients With EGFR-mutated Metastatic Non-small Cell Lung Cancer (NSCLC)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Apollomics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202104039
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase I Dose Level 1: APL-101 + Standard of Care Osimertinib (Experimental): * After 8-16 weeks of osimertinib, patients will be imaged as per standard of care. If imaging does not show disease progression, patients will continue on to study treatment with the combination of osimertinib and APL-101.
  * APL-101 is an oral drug which will be administered on an outpatient basis at the assigned dose twice daily on Days 1 through 28 of each 28-day cycle
  * Osimertinib is an oral drug which will be administered on an outpatient basis at a dose of 80 mg once daily on Days 1 through 28 of each 28-day cycle.
  Interventions: Drug: APL-101; Drug: Osimertinib
- Phase I Dose Level 2: APL-101 + Standard of Care Osimertinib (Experimental): * After 8-16 weeks of osimertinib, patients will be imaged as per standard of care. If imaging does not show disease progression, patients will continue on to study treatment with the combination of osimertinib and APL-101.
  * APL-101 is an oral drug which will be administered on an outpatient basis at the assigned dose twice daily on Days 1 through 28 of each 28-day cycle
  * Osimertinib is an oral drug which will be administered on an outpatient basis at a dose of 80 mg once daily on Days 1 through 28 of each 28-day cycle.
  Interventions: Drug: APL-101; Drug: Osimertinib
- Phase II: APL-101 + Standard of Care Osimertinib (Experimental): * After 8-16 weeks of osimertinib, patients will be imaged as per standard of care. If imaging does not show disease progression, patients will continue on to study treatment with the combination of osimertinib and APL-101.
  * APL-101 is an oral drug which will be administered on an outpatient basis at the assigned dose (this dose will be determined in Phase I of the study) twice daily on Days 1 through 28 of each 28-day cycle
  * Osimertinib is an oral drug which will be administered on an outpatient basis at a dose of 80 mg once daily on Days 1 through 28 of each 28-day cycle.
  Interventions: Drug: APL-101; Drug: Osimertinib

INTERVENTIONS:
Drug: APL-101 — -Provided by Apollomics
Drug: Osimertinib — -Given standard of care
  Other Names: Tagrisso

SUMMARY:
In this study, patients with metastatic non-small cell lung cancer that is EGFR-mutated, who have received at least 8 and not more than 12 weeks of treatment with osimertinib without demonstrating disease progression, will receive APL-101 in combination with osimertinib until progression. Dosing of APL-101 will be escalated until the maximum tolerated dose is determined, at which point 10 additional patients will be enrolled at that dose in the expansion cohort.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic non-small cell lung cancer, or locally advanced disease that is not amendable for curative intent therapy, with TKI-sensitive EGFR mutation through CLIA certified lab.
* Measurable disease by RECIST 1.1 with at least one lesion accessible for core biopsy.
* Planning to initiate treatment with standard of care osimertinib 80 mg QD. In order to continue treatment with osimertinib + APL-101, patients must have received at least 8 and no more than 16 weeks of SOC osimertinib without disease progression.
* At least 18 years of age.
* ECOG performance status ≤ 1
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Hemoglobin ≥ 9 g/dL (transfused Hgb allowed)
  * Total bilirubin ≤ 1.5 mg/dL or ≤ 26 µmol/L
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x institutional upper limit of normal (IULN) (≤ 5.0 x IULN if liver metastases)
  * Creatinine ≤2 x IULN or Creatinine clearance calculated by Cockcroft-Gault formula ≥60 ml/min
  * Serum calcium (after correcting for albumin level) ≤ IULN
  * Serum phosphorus ≤ IULN
* The effects of APL-101 on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study and for the duration of the study.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Prior treatment with osimertinib in the metastatic setting (outside of osimertinib given immediately prior to and during the enrollment period). Prior treatment with chemotherapy in the neoadjuvant, adjuvant, or first-line metastatic setting is however allowed.
* Prior immunotherapy and/or frontline EGFR-directed treatment in the metastatic setting. EGFR directed therapy in the adjuvant setting is permitted, as long as the disease-free interval between completion of adjuvant therapy with EGFR directed therapy and initiation of osimertinib is more than or equal to 1 year.
* Disease refractory to osimertinib, given immediately prior to and during enrollment period.
* A history of other malignancy with the exception of:

  * malignancies for which all treatment was completed at least 1 year before registration and the patient has no evidence of disease; or
  * known indolent malignancies, or malignancies that do not require active treatment and are unlikely not alter the course of treatment of metastatic NSCLC per treating physician.
* Currently receiving any other investigational agents or herbal medications
* Presence of symptomatic central nervous system metastases or neurologically unstable CNS symptoms (unable to taper steroids). Patients with treated brain metastases are eligible. Patients with asymptomatic brain metastases prior to initiation of osimertinib will be eligible to receive combination therapy as long as their disease is shown to be responsive to osimertinib.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to APL-101, osimertinib, or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, immune deficiencies, hepatitis B, untreated hepatitis C, uncontrolled diabetes, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, myocardial infraction within the past 6 months, uncontrolled cardiac arrhythmia, or prolonged QTc interval > 450 ms.
* Uncontrolled or symptomatic pleural or pericardial effusion. Effusion controlled by presence of an indwelling pleural catheter is not exclusionary.
* Decompensated heart failure or heart failure with reduced ejection fraction (<50%)
* Major surgery within 30 days prior to first day of study treatment (osimertinib + APL-101).
* Poorly controlled diarrheal or gastrointestinal disorders (grade 2 or higher diarrhea, nausea, or vomiting at baseline).
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Unresolved grade 2 or higher treatment-related toxicities (with the exception of endocrine abnormalities as a result of immunotherapies that are being managed with hormonal supplementation). However, if the treating physician is under the impression that the toxicity under question is unlikely to affect study participation, patient eligibility can be discussed with the PI on a subject by subject basis. After enrollment to this study, osimertinib-related toxicities must resolve to ≤ grade 1 before patient may begin combination therapy.
* Presence of interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Toxicity as measured by number of study treatment related adverse events (Phase I only) | Through 30 days after last dose of treatment (estimated to be 21 months)
  -Toxicity is measured by CTCAE v 5.0
Toxicity as measured by number of study discontinuations due to treatment-related adverse events (Phase I only) | Through 30 days after last dose of treatment (estimated to be 21 months)
  -Toxicity is measured by CTCAE v 5.0
Progression-free survival (PFS) (Phase II or received MTD only) | At 1 year
  * PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Patients who neither progress nor die by the data cutoff date will be censored at the last follow up date.
  * Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.

SECONDARY OUTCOMES:
Maximum tolerated dose of APL-101 (MTD) (Phase I only) | Through completion of cycle 1 (each cycle is 28 days) for all Phase I participants (estimated to be 19 months)
  * The maximum tolerated dose (MTD) is defined as the dose level immediately below the dose level at which 2 patients of a cohort (of 2 to 6 patients) experience dose-limiting toxicity during the first cycle.
Objective response rate as measured by the proportion of participants achieving a confirmed complete response or partial response (Phase II or received MTD only) | Through completion of treatment (estimated to be 20 months)
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumor marker level.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Duration of response (DOR) (Phase II or received MTD only) | Through completion of treatment (estimated to be 20 months)
  -Measured from the time measurement criteria are met for complete response, partial response or stable disease (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
Overall survival (OS) (Phase II or received MTD only) | Through 3 year follow-up (estimated to be 4 years and 8 months)
  -Overall survival (OS), defined as the duration of time from the start date of study treatment to death from any cause. Patients who are alive by the data cutoff date will be censored at the last follow up date.

CONTACTS AND LOCATIONS:
Overall Officials: Anjali Rohatgi, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu